CLINICAL TRIAL: NCT01298362
Title: Impact of Chemotherapy Followed by Aromatase Inhibitors on Bone Health of Women With ER-positive Early Breast Cancer in Real World Clinical Settings in Greece
Brief Title: Impact of Chemotherapy Followed by Aromatase Inhibitors on Bone Health of Women With ER-positive Early Breast Cancer
Acronym: POCHARBI
Status: Completed | Type: Observational
Sponsor: Hellenic Breast Surgeons Society (Other)
Responsible Party: Sponsor
Other Study IDs: POCHARBI - 2010/02
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Other Disorders of Bone Density and Structure
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AIs as first line therapy: Patients in postmenopausal status, with ER-positive early breast cancer, treated with an AI as first line therapy for 12 months.
  Interventions: Drug: Aromatase Inhibitors
- AIs after chemotherapy: Patients in postmenopausal status, with ER-positive early breast cancer, treated with an AI as maintenance therapy for 12 months after initial treatment with anthracycline- and/or taxane-based chemotherapy (chemotherapy treatment duration: 1-6 months).
  Interventions: Drug: Aromatase Inhibitors; Drug: Chemotherapy

INTERVENTIONS:
Drug: Aromatase Inhibitors
Drug: Chemotherapy
  Groups: AIs after chemotherapy

SUMMARY:
The purpose of this study is to identify the combined impact on bone loss as well as the incidence of bone fractures in women with estrogen receptor (ER)-positive, early breast cancer treated with an aromatase inhibitor (AI) either as first line therapy or as maintenance therapy after initial treatment with chemotherapy, in real life clinical settings in Greece.

DETAILED DESCRIPTION:
Subjects with ER-positive early breast cancer will be treated with AIs either as first line therapy or as maintenance therapy after initial treatment with chemotherapy. The total study duration will be 24 months comprising of a recruitment period of 12 months and a follow-up period of 12 months for each participating subject. The primary outcome variable is the mean percentage variation in lumbar spine (LS) bone mineral density (BMD) during the 12 month follow - up period. Measurements will be taken before and after chemotherapy and at the end of the 12 month follow - up period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Age ≥ 40 years.
* Female patients with ER-positive early breast cancer, who receive therapy with a third generation AI either as first line hormonal treatment or as maintenance therapy after first-line anthracycline- and/or taxane-based chemotherapy for a period no longer than 1 month (4 weeks) prior to inclusion in the present study.
* Women who have been rendered postmenopausal prior to chemotherapy commencement and at least 12 months from last menstrual period. For subjects who are amenorrheic for < 12 months (including patients who underwent hysterectomy, or received estrogen replacement therapy (ERT)/ hormone replacement therapy (HRT), they must have serum follicle stimulating hormone (FSH) ≥50 IU/L before the commencement of AI therapy.
* Patients with available data on lumbar spine and total hip bone mineral density (BMD) prior to chemotherapy initiation as well as before the commencement of AI therapy.

Exclusion Criteria:

* Prior administration of other endocrine therapy including tamoxifen.
* Chemotherapy-induced menopause.
* Evidence of diseases known to interfere with bone metabolism, such as hyperparathyroidism, hyperthyroidism, osteomalacia, chronic liver disease, renal failure, hypercortisolism, malabsorption, and immobilization.
* Evidence of bone metastasis or evidence of abnormal clinical laboratory parameters that are assessed as clinically significant by the investigator.
* Involvement in the planning and conduct of the study.
* Participation in other clinical study within a period of 3 months prior to any study related procedures.
* Patients with normal bone density or mild osteopenia (T score >= -2 in any site) under treatment with oral or intravenous bisphosphonates. Vitamin D and calcium supplements are allowed.
* Patients with severe osteopenia or osteoporosis (T score <= -2 in any site) under treatment with intravenous bisphosphonates. Oral bisphosphonates, Vitamin D and calcium supplements are allowed.
* Patients under treatment with oral or intravenous bisphosphonates before chemotherapy commencement.
* Patients that stopped hormone-replacement therapy (HRT) less than 3 months before chemotherapy commencement.
* Patients that received neo-adjuvant treatment.

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal female patients with ER-positive early breast cancer, who receive therapy with a third generation AI either as first line hormonal treatment or as maintenance therapy after first-line anthracycline- and/or taxane-based chemotherapy for a period no longer than 1 month (4 weeks) prior to inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos J Markopoulos, MD, MPhil, Principal Investigator — Associate Professor of Surgery-Athens University Medical School, Director of the Breast Unit-Athens Medical Centre Private Hospital
Locations (1):
- Hellenic Breast Surgeons Society, Athens, Attica, Greece

REFERENCES:
- [Derived] Markopoulos C, Koukouras D, Venizelos V, Karyda I, Xepapadakis G, Misitzis J, Kalogerakos K, Poulakaki F, Natsiopoulos J, Zobolas V, Savidou C, Antonopoulou Z, Tzoracoleftherakis E. Impact of chemotherapy followed by aromatase inhibitors on bone health of women with ER-positive early breast cancer in real world clinical settings in Greece: Results of the POCHARBI trial conducted by the Hellenic Society of Breast Surgeons. Breast. 2016 Jun;27:27-34. doi: 10.1016/j.breast.2016.02.007. Epub 2016 Mar 20. PMID 27212697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 290 post-menopausal female patients with ER-positive early breast cancer (BC) entered the study between February 2011 and December 2012. All 12 participating centers are hospitals where members of the Hellenic Society of Breast Surgeons operate.
Groups:
- CT Cohort: Patients were treated with a third generation AI, as subsequent endocrine therapy after initial treatment with chemotherapy (CT cohort), and were followed up for a 12-month period.
- HT Cohort: Patients were treated with a third generation AI, as adjuvant therapy (HT cohort) and were followed up for a 12-month period.
Period: Overall Study
Arm/Group | CT Cohort | HT Cohort
Started | 124 | 166
Completed | 86 | 123
Not Completed | 38 | 43
Not completed — Did not provide 12month BMD measurements | 38 | 43

BASELINE CHARACTERISTICS:
Population: This analysis is based on the 209 patients having full data (i.e. BMD measurements at baseline and at 12 months) however, their proﬁle is similar to the proﬁle of the whole sample of 290 patients originally enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | CT Cohort | HT Cohort | Total
Number analyzed (Participants) | 86 | 123 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 63 | 124
  >=65 years | 25 | 60 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.9) | 65.8 (9.2) | 63.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 123 | 209
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (5.4) | 29.3 (5.3) | 29.4 (5.3)
Smoker [Number; unit: participants]
  Current smoker | 20 | 21 | 41
  Ex smoker | 14 | 9 | 23
  Non smoker | 52 | 93 | 145
Physical Exercise [Number; unit: participants]
  Yes | 12 | 22 | 34
  No | 74 | 101 | 175
Osteopenia/osteoporosis before AI start [Number; unit: participants]
  Present | 16 | 34 | 50
  Absent | 70 | 89 | 159
1st degree relative with osteoporosis [Number; unit: participants]
  Yes | 7 | 15 | 22
  No | 79 | 108 | 187
Number of fractures in the past [Mean (Standard Deviation); unit: fractures] | 1.2 (0.4) | 1.2 (0.4) | 1.2 (0.4)
Fracture History [Number; unit: participants]
  Yes | 10 | 13 | 23
  No | 76 | 110 | 186
Orthopedic Surgery [Number; unit: participants]
  Yes | 5 | 9 | 14
  No | 81 | 114 | 195

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change in Lumbar Spine Bone Mineral Density From Baseline (Before Chemotherapy Commencement) to Month 12 of AI Therapy
Description: BMD was evaluated at lumbar spine (LS) and hip (HIP) with measurements taken before CT, before AI therapy and at the end of the 12 month followup period while on AI treatment. Dual Energy X-Ray Absorptiometry (DEXA scan) was used with all measurements performed with the Explorer absorptiometer produced by Hologic, Bedford, MA, USA in the same referral site in Athens, apart from two centres in other cities which used however the same absorptiometer model with identical software.
  The primary outcome variable was the mean percentage change in LS BMD between the pre CT treatment measurement and the post 12 months AI measurements in the CT cohort. The HT cohort was included as a control group.
Time Frame: Baseline and month 13-18 (1-6 months of chemotherapy + 12 months of AI therapy)
Population: Patients with LS BMd measurements both at baseline and at 12 months of AI therapy.
Measure: Mean (95% Confidence Interval); unit: percentage of change
Groups:
- HT Cohort: In the HT cohort patients were treated with a third generation AI, as adjuvant therapy (HT cohort) and were followed up for a 12-month period.
  The primary outcome variable was the mean percentage change in LS BMD between the pre CT treatment measurement and the post 12 months AI measurements in the CT cohort. The HT cohort was included as a control group.
  BMD measurements in HT cohort were taken before AI start and at 12 months.
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 86 | 0
percentage of change | -0.72 [-2.97 to 1.53] |

2. Secondary Outcome: Percentage Change in Total Hip Bone Mineral Density From Baseline to Month 12 of AI Therapy.
Time Frame: Baseline and month 13-18 (1-6 months of chemotherapy + 12 months of AI therapy)
Population: Patients with HIP BMD measurements both at baseline and at 12 months of AI therapy.
Measure: Mean (95% Confidence Interval); unit: percentage of change
Groups:
- HT Cohort: In the HT cohort patients were treated with a third generation AI, as adjuvant therapy (HT cohort) and were followed up for a 12-month period.
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 86 | 0
percentage of change | 0.83 [-2.56 to 4.23] |

3. Secondary Outcome: Percentage Change in Lumbar Spine Bone Mineral Density Before AI Commencement to Month 12 of Therapy for Patients Who Are Treated With AIs as First Line Therapy
Time Frame: From AI commencement to month 12 of AI therapy
Population: Patients with LS BMD measurements both at AI commencement and at 12 months of AI therapy.
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 0 | 123
percentage of change |  | 1.51 [-0.96 to 3.18]

4. Secondary Outcome: Percentage Change in Total Hip Bone Mineral Density Before AI Commencement to Month 12 of Therapy for Patients Who Are Treated With AIs as First Line Therapy
Time Frame: From AI commencement to month 12 of AI therapy
Population: Patients with HIP BMD measurements both at AI commencement and at 12 months of AI therapy.
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 0 | 123
percentage of change |  | -0.94 [-2.58 to 0.70]

5. Secondary Outcome: Bone Fracture Rate
Time Frame: During the 12 months of AI Therapy
Population: All patients with available 12 month follow-up during AI treatment
Measure: Number; unit: participants
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 86 | 123
participants | 0 | 0

6. Secondary Outcome: Mean Percentage Change in Lumbar Spine Bone Mineral Density From Baseline (Before Chemotherapy Commencement) to Chemotherapy Completion
Time Frame: Baseline and month 1-6 (depending on duration of chemotherapy)
Population: Patients with LS BMD measurements both at baseline (before chemotherapy commencement) and at chemotherapy completion
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 86 | 0
percentage of change | -0.19 [-2.12 to 1.74] |

7. Secondary Outcome: Mean Percentage Change in Lumbar Spine Bone Mineral Density From AI Commencement to Month 12 of Therapy.
Time Frame: Month 1-6 (depending on duration of chemotherapy) and month 13-18
Population: Patients with LS BMD measurements both at AI commencement and at 12 months of AI therapy.
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | CT Cohort | HT Cohort
Number analyzed (Participants) | 86 | 0
percentage of change | -0.59 [-3.18 to 2.00] |

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | CT Cohort | HT Cohort
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/123
Other Adverse Events (participants affected / at risk) | 0/86 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No